CLINICAL TRIAL: NCT03794583
Title: An Open-Label Extension Study of Inhaled Treprostinil in Patients With Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease (PH-COPD)
Brief Title: Inhaled Treprostinil in Participants With Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease (PH-COPD)
Acronym: PERFECT OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: United Therapeutics (Industry)
Collaborators: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PH-305
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Treprostinil; Lung Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Hypertension; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: This trial is not blinded. All participants will begin titration of study drug once all entry criteria have been met.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inhaled Treprostinil Solution (Experimental): Inhaled treprostinil solution (0.6 milligrams per milliliter [mg/mL], 6 mcg/breath) QID during waking hours.
  Interventions: Drug: Inhaled treprostinil solution

INTERVENTIONS:
Drug: Inhaled treprostinil solution — Inhaled treprostinil solution per dose and schedule specified in the arm

SUMMARY:
This open-label study will evaluate the safety of continued therapy with inhaled treprostinil in participants who have completed Study RIN-PH-304 (NCT03496623). This study hypothesizes that long-term safety findings will be similar to those observed in the randomized, placebo-controlled, double-blind, adaptive study 'A Phase 3, Randomized, Placebo-controlled, Double-blind, Adaptive Study to Evaluate the Safety and Efficacy of Inhaled Treprostinil in Patients with Pulmonary Hypertension due to Chronic Obstructive Pulmonary Disease (PH-COPD)(RIN-PH-304).

DETAILED DESCRIPTION:
This is a multi-center, open-label study for eligible participants who completed all scheduled study visits during the Treatment Period of Study RIN-PH-304.

Participants who provide informed consent for this open-label extension study on or prior to the final study visit of RIN-PH-304 may participate in the study, provided all other eligibility criteria are met. The RIN-PH-304 final study visit and the RIN-PH-305 Enrollment Visit will occur on the same day.

All participants will reinitiate inhaled treprostinil at 3 breathes (18 micrograms [mcg]) 4 times daily (QID) during waking hours. Study drug doses should be maximized to tolerability throughout the study, and dose titrations should occur as rapidly as possible (as directed by the Investigator) with a target dosing regimen of 15 breaths QID or the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Participant voluntarily gives informed consent to participate in the study.
2. Participant completed Study RIN-PH-304.
3. Women of childbearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must agree to practice abstinence or use 2 highly effective methods of contraception (defined as a method of birth control that results in a low failure rate, [less than 1% per year], such as approved hormonal contraceptives, barrier methods [such as condom or diaphragm] used with a spermicide, or an intrauterine device) for the duration of study treatment and for 48 hours after discontinuing study drug.
4. Males with a partner of childbearing potential must agree to use a barrier method (condom) with a spermicide for the duration of treatment and for at least 48 hours after discontinuing study drug.

Exclusion Criteria:

1. The participant is pregnant or lactating.
2. The participant was prematurely discontinued from Study RIN-PH-304.
3. The participant is intolerant to inhaled prostanoid therapy.
4. The participant is unwilling or unable to use Sponsor-provided devices (actigraph, spirometer, or smart device).
5. The participant is scheduled to receive another investigational drug, device, or therapy during the course of this study.
6. Any other clinically significant illness or abnormal laboratory value(s) that, in the opinion of the Investigator, might adversely affect the interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (27):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis Medical Center, Sacramento, California
  - St. Francis Sleep Allergy & Lung Institute, Clearwater, Florida
  - St. Vincent's Lung, Sleep, and Criticial Care Specialists, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - University of Illinois Medical Center, Chicago, Illinois
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Albany Medical Center, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Carl and Edyth Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Israel (3):
  - Lady Davis Carmel Medical Centre, Haifa
  - Hadassah-Hebrew University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tiva
- "Azienda Unita Sanitaria Locale Della Romagna Ospedale ""Gian Battista Morgagni"" - Luigi Pierantoni"" di Forli", Forlì, Forli, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 participants, who either successfully completed or were administratively terminated due to the COVID-19 pandemic from Study RIN-PH-304 (NCT03496623), chose to enroll in Study RIN-PH-305 (NCT03794583) open-label extension study.
Groups:
- Treprostinil: Participants received up to 90 micrograms (μg) of treprostinil for inhalation four times daily (QID), for up to 4 years
Period: Overall Study
Arm/Group | Treprostinil
Started | 41
Received At Least 1 Dose of Study Drug | 41
Completed | 0
Not Completed | 41
Not completed — Death | 8
Not completed — Study Terminated by Sponsor | 24
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of inhaled treprostinil.
Groups:
- Treprostinil: Participants received up to 90 μg of treprostinil for inhalation QID, for up to 4 years
Arm/Group | Treprostinil
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.24 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 31
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) can be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent was defined as any AE occurring/worsening at any time after a participant was exposed to study drug up until 7 days after the last dose of study drug. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to 4 years
Population: Safety population included all participants who received at least 1 dose of inhaled treprostinil.
Measure: Count of Participants; unit: Participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 41
Participants | 35

2. Secondary Outcome: Change From Baseline to Week 6 in 6-Minute Walk Distance (6MWD)
Description: 6MWD was calculated at peak exposure (10 to 60 minutes after dosing). 6-minute walk test (6MWT) was performed by standardized procedures for all participants. Participants were asked to walk a set course for 6 minutes (timed) and the distance walked (in meters) was recorded.
Time Frame: Baseline, Week 6
Population: All participants set included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants evaluable at the specified timeframe.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treprostinil
Number analyzed (Participants) | 38
meters
  Baseline | 226.5 (88.91)
  Change at Week 6: number analyzed (Participants) | 25
  Change at Week 6 | 15 (43.58)

3. Secondary Outcome: Change From Baseline to Week 6 in Borg Dyspnea Score
Description: The Borg Dyspnea Score was a 11-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (no dyspnea at all) to 10 (very, very severe dyspnea), with lower scores indicating less exertion (a better outcome). The Borg Dyspnea Score was to be evaluated immediately after the 6MWT.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treprostinil
Number analyzed (Participants) | 38
score on a scale
  Baseline | 5.03 (2.57)
  Change at Week 6: number analyzed (Participants) | 25
  Change at Week 6 | 0.38 (1.94)

4. Secondary Outcome: Change From Baseline to Week 6 in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: The NT-proBNP concentration is a biomarker associated with changes in right heart morphology and function. Improvement is defined as a decrease in the NT-proBNP plasma concentration.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram/liter (ng/L)
Arm/Group | Treprostinil
Number analyzed (Participants) | 40
nanogram/liter (ng/L)
  Baseline | 1279.6 (2080.19)
  Change at Week 6: number analyzed (Participants) | 29
  Change at Week 6 | -155.55 (558.96)

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Safety population included all participants who received at least 1 dose of inhaled treprostinil.
Arm/Group | Treprostinil
All-Cause Mortality (participants affected / at risk) | 8/41
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 22/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treprostinil (N=41)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Sudden death (General disorders) | 2
COVID-19 pneumonia (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treprostinil (N=41)
COVID-19 (Infections and infestations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4

LIMITATIONS AND CAVEATS:
Per sponsor decision, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03794583/Prot_SAP_000.pdf